CLINICAL TRIAL: NCT00911859
Title: A Randomized, Open-Label, Phase 2 Study of CNTO 328 (Anti-IL-6 Monoclonal Antibody) and VELCADE-Melphalan-Prednisone Compared With VELCADE-Melphalan-Prednisone for the Treatment of Previously Untreated Multiple Myeloma
Brief Title: A Study to Compare CNTO 328 (Anti-IL-6 Monoclonal Antibody) and VELCADE-Melphalan-Prednisone (VMP) With VMP Alone in Previously Untreated Multiple Myeloma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR015901; CNTO328MMY2001 (Other: Janssen Research & Development, LLC); 2008-007157-12 (EudraCT Number); NCT01710241 (obsolete NCT alias)
Record Dates: First submitted 2009-05-29; First posted 2009-06-02 (Estimated); Results first posted 2014-11-18 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; CNTO328; Interleukin-6 (IL-6); Monoclonal antibody; Anti-IL-6 monoclonal antibody; Bortezomib; Velcade; Melphalan; Prednisone
MeSH Terms: conditions — Multiple Myeloma | interventions — siltuximab; Bortezomib; Melphalan; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Part 1: VMP+Siltuximab 11 mg/kg (Experimental): Siltuximab 11 mg/kg as a 1-hour intravenous infusion every 3 weeks along with VMP (Velcade+Melphalan+Prednisone). Velcade 1.3 mg/m2 will be administered as an intravenous bolus injection according to the current approved package inserts. Melphalan 9 mg/m2 and prednisone 60 mg/m2 will be taken orally (by mouth).
  Interventions: Drug: Siltuximab11 mg/kg; Drug: Velcade (bortezomib); Drug: Melphalan; Drug: Prednisone
- Part 2, Arm A: VMP+Siltuximab 8.3 mg/kg or 11 mg/kg (Experimental): Siltuximab 8.3 mg/kg or 11 mg/kg as a 1-hour intravenous infusion every 3 weeks along with VMP. Velcade 1.3 mg/m2 will be administered as an intravenous bolus injection according to the current approved package inserts. Melphalan 9 mg/m2 and prednisone 60 mg/m2 will be taken orally
  Interventions: Drug: Siltuximab 8.3 mg/kg or 11 mg/kg; Drug: Velcade (bortezomib); Drug: Melphalan; Drug: Prednisone
- Part 2, Arm B: VMP (Active Comparator): Velcade 1.3 mg/m2 will be administered as an intravenous bolus injection according to the current approved package inserts. Melphalan 9 mg/m2 and prednisone 60 mg/m2 will be taken orally
  Interventions: Drug: Velcade (bortezomib); Drug: Melphalan; Drug: Prednisone

INTERVENTIONS:
Drug: Siltuximab11 mg/kg — Participants will receive siltuximab 11 mg/kg as a 1-hour intravenous infusion every 3 weeks in Part 1.
  Other Names: CNTO 328
  Arms: Part 1: VMP+Siltuximab 11 mg/kg
Drug: Siltuximab 8.3 mg/kg or 11 mg/kg — Participants will receive siltuximab 8.3 mg/kg or 11 mg/kg as a 1-hour intravenous infusion every 3 weeks for 9 cycles of treatment in Part 2, Arm A and in maintenance period.
  Other Names: CNTO 328
  Arms: Part 2, Arm A: VMP+Siltuximab 8.3 mg/kg or 11 mg/kg
Drug: Velcade (bortezomib) — Participants will receive Velcade 1.3 mg/m2 as an intravenous bolus injection according to the current approved package insert in Part 1.
  Other Names: bortezomib
  Arms: Part 1: VMP+Siltuximab 11 mg/kg
Drug: Velcade (bortezomib) — Participants will receive Velcade 1.3 mg/m2 as an intravenous bolus injection for 9 cycles of the treatment period in Part 2. It will be administered twice weekly for first 4 cycles (on Days 1, 4, 8, 11, 22, 25, 29, and 32, followed by a 10-day rest period) and once weekly for next 5 cycles (on Days 1, 8, 22, and 29, followed by a 13-day rest period)
  Other Names: bortezomib
  Arms: Part 2, Arm A: VMP+Siltuximab 8.3 mg/kg or 11 mg/kg
Drug: Melphalan — Participants will take melphalan 9 mg/m2 will be administered orally on Days 1 to 4, followed by a 38-day rest period in Part 1.
  Arms: Part 1: VMP+Siltuximab 11 mg/kg
Drug: Melphalan — Participants will receive melphalan according to currently approved package inserts. Melphalan 9 mg/m2 will be administered orally for 9 cycles of treatment period in Part 2, Arm A.
  Arms: Part 2, Arm A: VMP+Siltuximab 8.3 mg/kg or 11 mg/kg
Drug: Prednisone — Participants will take prednisone 60 mg/m2 will be administered orally on Days 1 to 4, followed by a 38-day rest period in Part 1.
  Arms: Part 1: VMP+Siltuximab 11 mg/kg
Drug: Prednisone — Participants will take prednisone 60 mg/m2 orally for 9 cycles of treatment period in Part 2, Arm A.
  Arms: Part 2, Arm A: VMP+Siltuximab 8.3 mg/kg or 11 mg/kg
Drug: Velcade (bortezomib) — Participants will receive Velcade 1.3 mg/m2 as an intravenous bolus injection according to the current approved package insert.
  Other Names: bortezomib
  Arms: Part 2, Arm B: VMP
Drug: Melphalan — Participants will take melphalan 9 mg/m2 orally according to currently approved package insert.
  Arms: Part 2, Arm B: VMP
Drug: Prednisone — Participants will take prednisone 60 mg/m2 orally according to the package insert.
  Arms: Part 2, Arm B: VMP

SUMMARY:
The purpose of this study is to evaluate safety and effectiveness of CNTO 328 (siltuximab) when it is administered together with velcade-melphalan-prednisone (VMP) in comparison with VMP alone in participants with multiple myeloma (a type of cancer that affects the blood and bone marrow).

DETAILED DESCRIPTION:
The study will be conducted in 2 parts (Part 1 and Part 2) and will consist of screening period up to 2 weeks; treatment period; maintenance period (CNTO 328 hereafter referred to as siltuximab) for a maximum of 18 months and follow up period until the study ends. Part 1 is an open-label (all people know the identity of the intervention), single group safety lead-in part to evaluate the safety of siltuximab. Approximately 12 patients will be treated with siltuximab in combination with VMP. If the safety profile of the combination is acceptable, the study will proceed to Part 2. Part 2 is a randomized (the study medication is assigned by chance), open-label, 2-arm (Arm A: siltuximab + VMP; Arm B: VMP alone) study. Approximately 104 patients will be equally randomized, followed by a maintenance period with siltuximab in particiants in Arm A who achieve a partial response (PR) or better. Particiants in both parts of the study will be treated up to a maximum of nine 6-week cycles provided there is no evidence of disease progression, unacceptable toxicity, or withdrawal from treatment. Study medication will be continued for at least 2 additional cycles after confirmation of complete response, and preferably for the full 9 cycles of the treatment period. Participants who will be receiving maintenance treatment after the 12-month effectiveness analysis may continue to receive treatment with siltuximab only after careful consideration by the treating physician and on evidence of clinical benefit and in the absence of unwarranted toxicities. Safety assessments will include evaluation of adverse events, clinical laboratory tests, eastern cooperative oncology group performance status, electrocardiogram, vital signs, and physical examination which will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of previously untreated multiple myeloma and not a candidate for high dose chemotherapy with stem cell transplantation
* Eastern cooperative oncology group performance status score of less than or equal to 2
* Measurable secretory disease, defined as either serum monoclonal paraprotein greater than or equal to 1 g/dL or urine monoclonal protein greater than 200 mg/24 hours
* Adequate laboratory results that will be confirmed by a study physician
* Agrees to protocol-defined use of effective contraception

Exclusion Criteria:

* Diagnosed with primary amyloidosis, asymptomatic or smoldering multiple myeloma or monoclonal gammopathy of undetermined significance
* Diagnosed with Waldenstrom's disease, or other conditions in which IgM M-protein is present in the absence of a clonal plasma cell infiltration with lytic bone lesions
* Received prior or current systemic therapy or stem cell transplantation for multiple myeloma
* Peripheral neuropathy or neuropathic pain (Grade 2 or higher)
* Received radiation therapy, plasmapheresis or surgery within 14 days
* Transplanted solid organ, with the exception of a corneal transplant
* Serious concurrent illness or history of uncontrolled heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2009-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development L.L.C Clinical Trial, Study Director — Janssen Research & Development L.L.C
Locations (37):
- United States (4):
  - Boston, Massachusetts
  - Chapel Hill, North Carolina
  - Philadelphia, Pennsylvania
  - Houston, Texas
- Australia (2):
  - Adelaide
  - Melbourne
- France (3):
  - Bordeaux
  - Montpellier
  - Strasbourg
- India (5):
  - Ahmedabad
  - Calicut
  - Hyderabad
  - Jaipur
  - Mumbai
- Israel (5):
  - Afula
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Ramat Gan
- Poland (5):
  - Bialystok
  - Chorzów
  - Gdynia
  - Lodz
  - Wroclaw
- Romania (3):
  - Baia Mare
  - Brasov
  - Iași
- Russia (4):
  - Arkhangelsk
  - Moscow
  - Nizhny Novgorod
  - Saint Petersburg
- Singapore, Singapore
- Seoul, South Korea
- Spain (4):
  - Barcelona
  - Madrid
  - Murcia
  - Salamanca

REFERENCES:
- [Derived] San-Miguel J, Blade J, Shpilberg O, Grosicki S, Maloisel F, Min CK, Polo Zarzuela M, Robak T, Prasad SV, Tee Goh Y, Laubach J, Spencer A, Mateos MV, Palumbo A, Puchalski T, Reddy M, Uhlar C, Qin X, van de Velde H, Xie H, Orlowski RZ. Phase 2 randomized study of bortezomib-melphalan-prednisone with or without siltuximab (anti-IL-6) in multiple myeloma. Blood. 2014 Jun 26;123(26):4136-42. doi: 10.1182/blood-2013-12-546374. Epub 2014 May 15. PMID 24833354

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 40 centers in 12 countries: Australia; France; India; Israel; Italy; Poland; Romania; Russian Federation; Singapore; South Korea; Spain; and the United States.
Pre-assignment Details: In Part 2, 105 participants received treatment (VMP: 53 and VMP+Siltuximab: 52). In the VMP+Siltuximab arm, 21 participants who achieved partial response or better entered the maintenance period and received only Siltuximab for 18 months, or until disease progression, unacceptable toxicity, or withdrawal from treatment, whichever occurred first.
Groups:
- Part 1: VMP + Siltuximab; Part 2: VMP + Siltuximab: Siltuximab 11 mg/kg as a 1-hour intravenous infusion every 3 weeks along with VMP. VMP: Velcade 1.3 mg/m2 was administered as an intravenous bolus injection according to the current approved package inserts. Melphalan 9 mg/m2 and prednisone 60 mg/m2 were taken orally.
- Part 2: VMP: Velcade 1.3 mg/m2 was administered as an intravenous bolus injection according to the current approved package inserts. Melphalan 9 mg/m2 and prednisone 60 mg/m2 were taken orally.
Period: Treatment Period
Arm/Group | Part 1: VMP + Siltuximab | Part 2: VMP | Part 2: VMP + Siltuximab
Started | 12 | 54 | 52
Received Treatment | 12 | 53 | 52
Completed | 4 | 33 | 27
Not Completed | 8 | 21 | 25
Not completed — Adverse Event | 3 | 3 | 7
Not completed — Death | 1 | 3 | 5
Not completed — Lack of Efficacy | 1 | 7 | 5
Not completed — Physician Decision | 3 | 3 | 3
Not completed — Withdrawal by Subject | 0 | 4 | 5
Not completed — Did not receive study treatment | 0 | 1 | 0
Period: Maintainance Period
Arm/Group | Part 1: VMP + Siltuximab | Part 2: VMP | Part 2: VMP + Siltuximab
Started | 0 | 0 | 21 (Participants who received siltuximab only during the 18-month maintenance period)
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 21
Not completed — Lack of Efficacy | 0 | 0 | 9
Not completed — Physician Decision | 0 | 0 | 9
Not completed — Withdrawal by Subject | 0 | 0 | 3
Period: Follow-up Period
Arm/Group | Part 1: VMP + Siltuximab | Part 2: VMP | Part 2: VMP + Siltuximab
Started | 12 (Participants followed until death or 3.5 years after the last participant was assigned to treatment) | 53 (Participants followed until death or 3.5 years after the last participant was assigned to treatment) | 52 (Participants followed until death or 3.5 years after the last participant was assigned to treatment)
Completed | 1 | 7 | 11
Not Completed | 11 | 46 | 41
Not completed — Death | 5 | 8 | 10
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 4
Not completed — Study terminated by sponsor | 5 | 33 | 27

BASELINE CHARACTERISTICS:
Groups:
- Part 1: VMP (Velcade+Melphalan+Prednisone) + Siltuximab; Part 2: VMP (Velcade+Melphalan+Prednisone) + Siltuximab: Siltuximab 11 mg/kg as a 1-hour intravenous infusion every 3 weeks along with VMP. VMP: Velcade 1.3 mg/m2 was administered as an intravenous bolus injection according to the current approved package inserts. Melphalan 9 mg/m2 and prednisone 60 mg/m2 were taken orally.
- Part 2: VMP (Velcade+Melphalan+Prednisone): Velcade 1.3 mg/m2 was administered as an intravenous bolus injection according to the current approved package inserts. Melphalan 9 mg/m2 and prednisone 60 mg/m2 were taken orally.
- Total: Total of all reporting groups
Arm/Group | Part 1: VMP (Velcade+Melphalan+Prednisone) + Siltuximab | Part 2: VMP (Velcade+Melphalan+Prednisone) | Part 2: VMP (Velcade+Melphalan+Prednisone) + Siltuximab | Total
Number analyzed (Participants) | 12 | 54 | 52 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.6 (6.3) | 70.3 (7.27) | 71.6 (4.76) | 71.2 (6.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 30 | 29 | 66
  Male | 5 | 24 | 23 | 52
Region of Enrollment [Number; unit: participants]
  AUSTRALIA | 0 | 2 | 2 | 4
  FRANCE | 0 | 5 | 2 | 7
  INDIA | 0 | 3 | 1 | 4
  ISRAEL | 0 | 7 | 5 | 12
  ITALY | 0 | 2 | 2 | 4
  POLAND | 0 | 5 | 11 | 16
  ROMANIA | 0 | 2 | 0 | 2
  RUSSIAN FEDERATION | 0 | 10 | 10 | 20
  SINGAPORE | 0 | 3 | 2 | 5
  SOUTH KOREA | 0 | 7 | 8 | 15
  SPAIN | 12 | 5 | 7 | 24
  UNITED STATES | 0 | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Complete Response (CR) - European Group for Blood and Marrow Transplantation (EBMT) Criteria
Description: CR was assessed using EMBT criteria: disappearance of the original monoclonal paraprotein from the blood and urine on at least 2 determinations for a minimum of 6 weeks by immunofixation studies, <5% plasma cells in the bone marrow on at least 1 determination, if skeletal survey is available: no increase in the size or number of lytic bone lesions (development of a compression fracture does not exclude response), disappearance of soft tissue plasmacytomas for at least 6 weeks.
Time Frame: Up to disease progression, approximately 3 years
Population: Response-evaluable population: Participants who had a confirmed diagnosis of multiple myeloma and measurable disease according to the EBMT criteria were evaluated for disease response. Also, participants must have received at least 1 administration of study medication and have at least 1 post-baseline disease assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2: VMP (Velcade+Melphalan+Prednisone) | Part 2: VMP (Velcade+Melphalan+Prednisone) + Siltuximab
Number analyzed (Participants) | 49 | 49
Percentage of participants | 22.4 | 26.5

2. Secondary Outcome: Percentage of Participants Who Achieved Overall Response ie, Complete Response (CR) or Partial Response (PR) - European Group for Blood and Marrow Transplantation (EBMT) Criteria
Description: CR or PR was assessed using EBMT criteria. CR: disappearance of the original monoclonal paraprotein from the blood and urine on at least 2 determinations for a minimum of 6 weeks by immunofixation studies, <5% plasma cells in the bone marrow on at least 1 determination, if skeletal survey is available: no increase in the size or number of lytic bone lesions (development of a compression fracture does not exclude response), disappearance of soft tissue plasmacytomas for at least 6 weeks; PR: >=50% reduction in the level of serum monoclonal paraprotein for at least 2 determinations 6 weeks apart, if present, reduction in 24-hour urinary light chain excretion by either >=90% or to <200 mg for at least 2 determinations 6 weeks apart, >=50% reduction in the size of soft tissue plasmacytomas (by clinical or radiographic examination) for at least 6 weeks, if skeletal survey is available: no increase in size or number of lytic bone lesions
Time Frame: Up to disease progression, approximately 3 years
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2: VMP (Velcade+Melphalan+Prednisone) | Part 2: VMP (Velcade+Melphalan+Prednisone) + Siltuximab
Number analyzed (Participants) | 49 | 49
Percentage of participants | 79.6 | 87.8

3. Secondary Outcome: Percentage of Participants Who Achieved Stringent Complete Response (sCR) - International Myeloma Working Group (IMWG) Criteria
Description: sCR was assesses by IMWG Criteria: Negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas, <=5% plasma cells in bone marrow, normal free light chain ratio, absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence. sCR is a CR that has been confirmed by immunofixation + free light chain assay + either bone marrow immunohistochemistry or immunofluorescence
Time Frame: Up to disease progression, approximately 3 years
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2: VMP (Velcade+Melphalan+Prednisone) | Part 2: VMP (Velcade+Melphalan+Prednisone) + Siltuximab
Number analyzed (Participants) | 49 | 49
Percentage of participants | 6.1 | 4.1

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time between randomization and either disease progression or death, whichever occurred first.
Time Frame: From the date of randomization until disease progression or death, whichever occurred first, as assessed up to the last efficacy assessment for disease progression (approximately 3 years)
Population: Intent-to-treat (ITT) population: all randomized participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 2: VMP (Velcade+Melphalan+Prednisone) | Part 2: VMP (Velcade+Melphalan+Prednisone) + Siltuximab
Number analyzed (Participants) | 54 | 52
Days | 518 [460 to 582] | 519 [443 to 673]

5. Secondary Outcome: 1-year Progression-Free Survival (PFS) Rate
Description: The 1-year PFS rate was defined as the percentage of participants surviving 1 year after randomization without disease progression or death.
Time Frame: 1 year
Population: Intent-to-treat (ITT) population: all randomized participants
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2: VMP (Velcade+Melphalan+Prednisone) | Part 2: VMP (Velcade+Melphalan+Prednisone) + Siltuximab
Number analyzed (Participants) | 54 | 52
Percentage of participants | 77.5 | 72.1

6. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as length from the earliest date a participant achieved a complete response (CR) or partial response (PR) to either date for disease progression (including relapse from CR) or the censoring date for progressive disease. Responders without disease progression were censored at the last efficacy assessment for disease progression.
Time Frame: From the date participants achieved CR or PR to either date for disease progression (including relapse from CR) or the censoring date for progressive disease, as assessed Up to 30 days after last dose of study medication
Population: Included participants in the randomized population who achieved CR or PR.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 2: VMP (Velcade+Melphalan+Prednisone) | Part 2: VMP (Velcade+Melphalan+Prednisone) + Siltuximab
Number analyzed (Participants) | 39 | 43
Days | 497 [457 to 637] | 583 [449 to NA] — Insufficient number of participants with events; therefore, upper limit of 95% CI not reached.

7. Secondary Outcome: 1-year Survival Rate
Description: Percentage of participants who are alive at the end of year 1 after randomization
Time Frame: 1 year
Population: Intent-to-treat (ITT) population: all randomized participants
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2: VMP (Velcade+Melphalan+Prednisone) | Part 2: VMP (Velcade+Melphalan+Prednisone) + Siltuximab
Number analyzed (Participants) | 54 | 52
Percentage of participants | 87.8 | 87.5

8. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time interval in days between the date of randomization and the participant's death from any cause.
Time Frame: From the date of randomization till the date of death, as assessed up to the end of study (approximately 3 years)
Population: Intent-to-treat (ITT) population: all randomized participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 2: VMP (Velcade+Melphalan+Prednisone) | Part 2: VMP (Velcade+Melphalan+Prednisone) + Siltuximab
Number analyzed (Participants) | 54 | 52
Days | NA [NA to NA] — Insufficient number of participants with events; therefore, median and 95% CI not reached. | NA [783 to NA] — Insufficient number of participants with events; therefore, median and upper limit of 95% CI not reached.

9. Secondary Outcome: Change From Baseline to Cycle 9 in Global Health Status/Quality of Life Subscale of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ C30)
Description: Global health status/quality of life is a subscale of the EORTC QOL C30, which comprises two questions related to overall health/quality of life during the past week. The raw score to each question ranged from 1 (very poor) to 7 (excellent). The raw mean score of health status/quality of life subscale is calculated for each participant and a linear transformation applied to standardize the raw score, so that scores range from 0 to 100; a higher score represents a higher ("better") health and quality of life.
Time Frame: Baseline (Day 1 predose) and Cycle 9 (Week 54)
Population: Intent-to-treat (ITT) population: all randomized participants with evaluable data during baseline and Cycle 9
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Part 2: VMP (Velcade+Melphalan+Prednisone) | Part 2: VMP (Velcade+Melphalan+Prednisone) + Siltuximab
Number analyzed (Participants) | 31 | 25
Scores on a scale | 14.78 (25.250) | 8.33 (31.088)

ADVERSE EVENTS:
Time Frame: Up to 30 days after the last dose of study medication
Description: For Safety analyses all randomized participants who received at least 1 dose of study agents were analyzed. Data are presented for 117 participants in the treatment period (Part 1 and Part 2) and 21 participants who entered maintenance period (after achieving partial response or better in the Part 2 treatment period while receiving VPM+siltuximab)
Groups:
- Part 2, Maintenance Period: Siltuximab: Siltuximab 8.3 mg/kg or 11 mg/kg as a 1-hour intravenous infusion every 3 weeks, during the maintenance period
Arm/Group | Part 1: VMP (Velcade+Melphalan+Prednisone) + Siltuximab | Part 2: VMP (Velcade+Melphalan+Prednisone) | Part 2: VMP (Velcade+Melphalan+Prednisone) + Siltuximab | Part 2, Maintenance Period: Siltuximab
Serious Adverse Events (participants affected / at risk) | 8/12 | 27/53 | 30/52 | 1/21
Other Adverse Events (participants affected / at risk) | 12/12 | 51/53 | 51/52 | 15/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: VMP (Velcade+Melphalan+Prednisone) + Siltuximab (N=12) | Part 2: VMP (Velcade+Melphalan+Prednisone) (N=53) | Part 2: VMP (Velcade+Melphalan+Prednisone) + Siltuximab (N=52) | Part 2, Maintenance Period: Siltuximab (N=21)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac Failure (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac Failure Acute (Cardiac disorders) | 0 | 0 | 1 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Steroid Withdrawal Syndrome (Endocrine disorders) | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus Paralytic (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Adverse Drug Reaction (General disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 3 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis Escherichia Coli (Infections and infestations) | 0 | 1 | 0 | 0
H1n1 Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Hepatitis B (Infections and infestations) | 1 | 0 | 0 | 0
Lobar Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Parotitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 3 | 5 | 7 | 0
Pneumonia Pneumococcal (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 1 | 0
Septic Shock (Infections and infestations) | 1 | 1 | 0 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Weight Decreased (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Bone Lesion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Adenocarcinoma Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Multiple Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cerebral Ischaemia (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoglycaemic Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Lacunar Infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Metabolic Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 2 | 0
Completed Suicide (Psychiatric disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 1 | 3 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 1 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 2 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Status Asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Leukocytoclastic Vasculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 2 | 0 | 0
Hypovolaemic Shock (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: VMP (Velcade+Melphalan+Prednisone) + Siltuximab (N=12) | Part 2: VMP (Velcade+Melphalan+Prednisone) (N=53) | Part 2: VMP (Velcade+Melphalan+Prednisone) + Siltuximab (N=52) | Part 2, Maintenance Period: Siltuximab (N=21)
Anaemia (Blood and lymphatic system disorders) | 5 | 19 | 12 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 5 | 6 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 3 | 4 | 0
Neutropenia (Blood and lymphatic system disorders) | 11 | 25 | 34 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 21 | 30 | 5
Atrial Fibrillation (Cardiac disorders) | 1 | 2 | 2 | 0
Conjunctivitis (Eye disorders) | 0 | 2 | 4 | 0
Dry Eye (Eye disorders) | 0 | 4 | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 3 | 2 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 2 | 3 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 6 | 4 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 4 | 4 | 0
Constipation (Gastrointestinal disorders) | 8 | 16 | 18 | 2
Diarrhoea (Gastrointestinal disorders) | 7 | 21 | 18 | 2
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 4 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 6 | 3 | 1
Gastritis (Gastrointestinal disorders) | 0 | 3 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 2 | 4 | 0
Mouth Ulceration (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 4 | 21 | 16 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 15 | 12 | 1
Asthenia (General disorders) | 10 | 18 | 10 | 0
Chest Pain (General disorders) | 0 | 5 | 6 | 1
Chills (General disorders) | 1 | 3 | 3 | 0
Fatigue (General disorders) | 0 | 8 | 12 | 2
Malaise (General disorders) | 1 | 3 | 0 | 0
Mucosal Discolouration (General disorders) | 1 | 0 | 0 | 0
Oedema (General disorders) | 2 | 4 | 0 | 0
Oedema Peripheral (General disorders) | 3 | 4 | 16 | 0
Pain (General disorders) | 0 | 2 | 3 | 1
Pyrexia (General disorders) | 1 | 15 | 9 | 0
Spinal Pain (General disorders) | 1 | 0 | 0 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 2 | 6 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 5 | 6 | 0
H1n1 Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 3 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 5 | 4 | 2
Nipple Infection (Infections and infestations) | 1 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 1 | 0 | 0 | 0
Oral Candidiasis (Infections and infestations) | 3 | 3 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 1 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 2 | 1 | 3 | 0
Respiratory Tract Infection Viral (Infections and infestations) | 0 | 3 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 3 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 6 | 5 | 2
Urinary Tract Infection (Infections and infestations) | 1 | 2 | 5 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Weight Decreased (Investigations) | 0 | 6 | 6 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 4 | 18 | 9 | 1
Enzyme Abnormality (Metabolism and nutrition disorders) | 0 | 1 | 4 | 0
Fluid Retention (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 2 | 3 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 2 | 7 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 4 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 4 | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 6 | 6 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 7 | 9 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 6 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 4 | 3 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 4 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 2 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 7 | 10 | 3
Dizziness (Nervous system disorders) | 2 | 9 | 11 | 1
Essential Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 3 | 4 | 1
Monoparesis (Nervous system disorders) | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 5 | 16 | 10 | 0
Paraesthesia (Nervous system disorders) | 0 | 4 | 4 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 9 | 34 | 31 | 1
Somnolence (Nervous system disorders) | 1 | 2 | 1 | 0
Syncope (Nervous system disorders) | 0 | 3 | 2 | 0
Tremor (Nervous system disorders) | 1 | 1 | 1 | 0
Agitation (Psychiatric disorders) | 1 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 5 | 4 | 0
Confusional State (Psychiatric disorders) | 0 | 3 | 1 | 0
Depression (Psychiatric disorders) | 2 | 3 | 3 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 3 | 13 | 10 | 1
Dysuria (Renal and urinary disorders) | 0 | 2 | 4 | 0
Renal Impairment (Renal and urinary disorders) | 0 | 1 | 6 | 0
Pelvic Pain (Reproductive system and breast disorders) | 0 | 0 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 10 | 11 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 8 | 6 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 4 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 5 | 5 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 4 | 7 | 0
Scar (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 7 | 4 | 0
Hypotension (Vascular disorders) | 1 | 2 | 7 | 1
Orthostatic Hypotension (Vascular disorders) | 2 | 2 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days